CLINICAL TRIAL: NCT01067677
Title: Rescue Emetic Therapy for Children Having Elective Therapy
Brief Title: Rescue Emetic Therapy for Children Having Elective Surgery
Acronym: RETCHES
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We do not have the funding or resources to complete the study at this time
Sponsor: Franklyn Cladis (Other)
Responsible Party: Sponsor-Investigator, Franklyn Cladis, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-Cladis
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Post Operative Nausea and Vomiting; Rescue Emetic Therapy
Keywords: PONV; Post operative nausea and vomiting; rescue emetic therapy
MeSH Terms: conditions — Vomiting; Postoperative Nausea and Vomiting | interventions — Metoclopramide; Ondansetron; Diphenhydramine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Metoclopramide (Experimental): rescue emetic therapy
  Interventions: Drug: Metaclopramide
- Ondansetron (Experimental): Rescue emetic therapy
  Interventions: Drug: Ondansetron
- Diphenhydramine (Experimental): Rescue emetic therapy
  Interventions: Drug: diphenhydramine
- Saline (Placebo Comparator): Placebo
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Metaclopramide — 0.5 mg/kg for rescue after PONV
  Arms: Metoclopramide
Drug: Ondansetron — 0.1 mg/kg (max 4 mg0
  Arms: Ondansetron
Drug: diphenhydramine — 0.25 mg/kg (max 25 mg)
  Arms: Diphenhydramine
Drug: Saline — equal volume (5 ml)as experimental rescue medications
  Arms: Saline

SUMMARY:
To compare ondansetron, metoclopramide, diphenhydramine, and placebo in order to determine which anti-emetic is most efficacious as a "rescue therapy" for pediatric patients ages 3-18 who have post-operative vomiting after a standardized prophylactic regimen of ondansetron and dexamethasone. We hypothesize that anti-emetics with a different mechanism of action than the prophylactic regimen will be the most effective "rescue therapy" in children having surgery in an ambulatory surgery center.

1. Problem: Despite commonly-used anti-emetics for prophylaxis, some children still go on to develop post-operative vomiting (POV).

   Goal: To determine which anti-emetic--ondansetron, metoclopramide, diphenhydramine, or placebo--is most efficacious for pediatric patients in this situation.
2. Hypothesis: Anti-emetic medications that have a different mechanism of action than the prophylactic regimen will be the most efficacious "rescue therapy."
3. Hypothesis: Metoclopramide at the dose of 0.5 mg/kg (max dose 20 mg) will be more effective than ondansetron, diphenhydramine, or placebo as "rescue therapy."

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients 3-17 years old
2. Patients scheduled for tonsillectomy and/or adenoidectomy (with and without myringotomy) , or dental restoration,
3. Patients receiving a general anesthetic (inhaled agent without nitrous oxide) with POV prophylaxis with two agents (ondansetron and dexamethasone)
4. Post operative vomiting in PACU or second stage recovery requiring antiemetic rescue.

Exclusion Criteria:

1. Vomiting in the past 24 hours or antiemetics in previous 24 hours
2. Allergy or sensitivity to ondansetron, dexamethasone, metoclopramide, or diphenhydramine
3. Patients with diabetes
4. Patients with seizures
5. Patients receiving a benzodiazepine premedication

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Primary-Incidence of POV after rescue antiemetic in PACU, car ride home, day of surgery, and POD #1 and 2 | 48 hrs

SECONDARY OUTCOMES:
Secondary - a. Discharge times | 48 hrs
Adverse events (headaches, sedation, dystonic reaction, dry mouth) | 48 hrs
POV risk factors. age, personal or family history of PONV, history of motion sickness, personal or family history of smoking | 48 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Franklyn P Cladis, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- The Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States